CLINICAL TRIAL: NCT03805243
Title: Evaluation of the Signals électrophysiologiques Measured by Intelligent Textiles
Brief Title: Evaluation of the Signals Electrophysiological Measured by Intelligent Textiles
Acronym: DATASET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of products design
Sponsor: BioSerenity (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A02535-48
Record Dates: First submitted 2018-04-23; First posted 2019-01-15 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: All subject would likely test each the 5 devices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- test of sensors for somnonaute device (Experimental): monitoring with sensors
  Interventions: Device: test of sensors for somnonaute device
- test of sensors for uronaute device (Experimental): monitoring with sensors
  Interventions: Device: test of sensors for uronaute device
- test of sensors for toconaute device (Experimental): monitoring with sensors
  Interventions: Device: test of sensors for toconaute device
- test of sensors for cardioskin device (Experimental): monitoring with sensors
  Interventions: Device: test of sensors for cardioskin device
- test of sensors for neuronaute device (Experimental): monitoring with sensors
  Interventions: Device: test of sensors for neuronaute device

INTERVENTIONS:
Device: test of sensors for somnonaute device — test of sensors
  Arms: test of sensors for somnonaute device
Device: test of sensors for uronaute device — test of sensors
  Arms: test of sensors for uronaute device
Device: test of sensors for toconaute device — test of sensors
  Arms: test of sensors for toconaute device
Device: test of sensors for neuronaute device — test of sensors
  Arms: test of sensors for neuronaute device
Device: test of sensors for cardioskin device — test of sensors
  Arms: test of sensors for cardioskin device

SUMMARY:
BioSerenity suggests developing innovative solutions, from intelligent clothes which can be used in a hospital environment or at home. These textiles allow, in particular, to measure the biophysiological signals while letting to the participant the freedom pursue its daily activities.

BioSerenity has already developed two wearable wireless and portable medical devices: cardioskin with textile ECG electrods , and the Neuronaute with textile EEG, EMG electrods.

The aim of the study is to test these sensors to optimize their signal to integrate them in future Bioserenity devices like a somnonaute to help diagnosis of sleep disorders, like uronaute to help diagnosis of urination disorders, like toconaute to help monitoring of pregnancy. Others CE-marked sensors developed by others manufacturers will be tested to choose those that will be integrated in the Bioserenity devices.

DETAILED DESCRIPTION:
The various alone sensors tested in the clinical trial (sensors of Bioserenity and the other manufacturers), will supply information which will allow to develop future devices. Some of these sensors will then be selected to integrate them.

The tests will be made according to the therapeutic area of the concerned device(plan). There are 5 therapeutic areas:

Cardiovascular (Cardioskin device), neurology ( Neuronaute device), urology ( Uronaute device), obstetrics ( Toconaute device), somnologie (Somnonaute device).

One subject would likely test either one sensor of a device or multiple sensors, either an entire device.

ELIGIBILITY:
Inclusion Criteria:

* women or men >18 years
* affiliation to a social security system

Exclusion Criteria:

* Wounds or wounds on the body and the scalp;
* Refusal of consent, minor
* Not membership to the Social Security
* Participant not capable of following the procedure of use (according to the judgment of the investigator);
* Brain surgery that took place less than a week ago
* Allergy known about the money, the polyamide, the silicone, the synthetic materials;
* Sensory Disorders(Confusions) returning the insensible subject to the pain;
* Motor or mental disorders preventing the subject from expressing his pain;
* Behavioral problems that make the subject excessively agitated or aggressive;
* People with cardio-respiratory problems likely to be aggravated by the slight compression of the thorax;
* Subject equipped with an electrical stimulation device;
* Unsuitable anthropometric Parameters (for the women, the sizes superior to 24 will be excluded and for the men(people) those superior to 34);
* Pregnancy clinically detectable or known for the subject;
* Current(in class) Participation in a clinical trial or participation in a previous clinical trial understanding(including) a period of not past(over) deficiency at the time of this clinical trial.
* Predisposition in the headaches of tension (the compression exercised by the hat(cap) can activate(start) in certain cases a headache);
* Use of the device(plan) within the framework of a resuscitation or of intensive care;
* Participating carrier of a defibrillator, a stimulating of the vagus nerve, or quite different surgical high-frequency device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Sensor quality validation | 24 months
  Signal is considered as of "good quality" " not good quality" regarding criteria of signal patterns : eg amplitude of signal, regularity..

CONTACTS AND LOCATIONS:
Overall Officials: quang TRAN, Study Director — BioSerenity
Locations (1):
- Institut Du Cerveau Et de La Moelle Epiniere, Paris, France

IPD SHARING:
Plan to Share IPD: No